CLINICAL TRIAL: NCT02746224
Title: Reconstruction Techniques and Vascular Approach After Laparoscopic Left Hemicolectomy and Laparoscopic Low Anterior Resection for Rectal Cancer: a Randomized Clinical Trial
Brief Title: Reconstruction Techniques and Vascular Approach After Laparoscopic Left Hemicolectomy and Rectum Low Anterior Resection
Acronym: TAHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Pere Planellas Giné, MD-PhD, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34502
Record Dates: First submitted 2016-04-13; First posted 2016-04-21 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Rectal Tumors
Keywords: Colorectal cancer; Colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- group 1A (Other): the surgical technique initially dissects the inferior mesenteric vein (IMV).
  Interventions: Procedure: Initially dissection of inferior mesenteric vein
- group 1B (Other): the surgical technique initially dissects the inferior mesenteric artery (IMA).
  Interventions: Procedure: Initially dissection of inferior mesenteric artery
- group 2A (Other): the patients will have a latero-terminal colorectal anastomosis
  Interventions: Procedure: Initially dissection of inferior mesenteric vein; Procedure: Latero-terminal colorectal anastomosis
- group 2B (Other): the patients will have a termino-terminal colorectal anastomosis.
  Interventions: Procedure: Initially dissection of inferior mesenteric artery; Procedure: Termino-terminal colorectal anastomosis

INTERVENTIONS:
Procedure: Initially dissection of inferior mesenteric vein — Laparoscopic left hemicolectomy for left colon cancer or laparoscopic low anterior resection for rectal cancer. In the group 1A the surgical technique initially dissects the inferior mesenteric vein (IMV)
  Arms: group 1A; group 2A
Procedure: Initially dissection of inferior mesenteric artery — Laparoscopic left hemicolectomy for left colon cancer or laparoscopic low anterior resection for rectal cancer. In the group 1B the surgical technique initially dissects the inferior mesenteric artery.
  Arms: group 1B; group 2B
Procedure: Latero-terminal colorectal anastomosis — The patients who will undergo a colorectal anastomosis will be included in the study 2 and will be randomized to group 2A and group 2B: in group 2A the patients will have a latero-terminal colorectal anastomosis and in group 2B a termino-terminal colorectal anastomosis.
  Arms: group 2A
Procedure: Termino-terminal colorectal anastomosis — The patients who will undergo a colorectal anastomosis will be included in the study 2 and will be randomized to group 2A and group 2B: in group 2A the patients will have a latero-terminal colorectal anastomosis and in group 2B a termino-terminal colorectal anastomosis.
  Arms: group 2B

SUMMARY:
This is an interventional, controlled and randomized single-center clinical trial with patients diagnosed with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer.

All patients included in the study (study 1) are randomized into two groups (group 1A and group 1B): in the group 1A the surgical technique initially dissects the inferior mesenteric vein (IMV) and in the group 1B the surgical technique initially dissects the inferior mesenteric artery.

The patients who will undergo a colorectal anastomosis will be included in the study 2 and will be randomized to group 2A and group 2B: in group 2A the patients will have a latero-terminal colorectal anastomosis and in group 2B a termino-terminal colorectal anastomosis.

Study hypothesis:

Study 1: the surgical technique that initially dissects the IMV presents a greater number of total resected lymph nodes compared to the technique that initially dissects the IMA.

Study 2: latero-terminal anorectal anastomosis has a better anorectal functional outcome than termino-terminal anorectal anastomosis.

Primary outcome measures:

* Study 1:To compare the total number of resected lymph nodes and the distance to the surgical margins between the two arms (1A and 1B).
* Study 2: to compare the anorectal functional outcome at 12 months after surgery or ileostomy closure between the two arms (2A and 2B). The anorectal function will be assessed by the scores of the validated Colorectal Functional Outcome Questionnaire (COREFO) and the validated scale LARS (Syndrome anterior resection of the rectum).

Secondary outcome measures:

* Study 1: to compare the duration of surgery, bleeding and need for surgical conversion between the two arms (1A and 1B). Another objectives are to compare the incidence of postoperative complications (measured by the Clavien-Dindo classification) and survival.
* Study 2: to compare the quality of life and anorectal functional outcomes at : 6, 12, 18 and 24 months after intervention (or ileostomy closure) between the two arms (2A and 2B). The anorectal function will be assessed by the validated COREFO questionnaire and the LARS scale. The quality of life will be assessed by the validated questionnaire of quality of life: SF-36. Another objective is to compare the incidence of postoperative complications assessed by the Clavien-Dindo classification and the incidence of anastomotic leakage.

DETAILED DESCRIPTION:
This is an interventional, controlled and randomized single-center clinical trial with patients diagnosed with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer.

Methods:

All patients included in the study (study 1) are randomized into two groups (group 1A and group 1B): in the group 1A the surgical technique initially dissects the inferior mesenteric vein (IMV) and in the group 1B the surgical technique initially dissects the inferior mesenteric artery.

The patients who will undergo a colorectal anastomosis will be included in the study 2 and will be randomized to group 2A and group 2B: in group 2A the patients will have a latero-terminal colorectal anastomosis and in group 2B a termino-terminal colorectal anastomosis.

Study hypothesis:

Study 1: the surgical technique that initially dissects the IMV presents a greater number of total resected lymph nodes compared to the technique that initially dissects the IMA.

Study 2: latero-terminal anorectal anastomosis has a better anorectal functional outcome than termino-terminal anorectal anastomosis.

Primary outcome measures:

* Study 1:To compare the total number of resected lymph nodes and the distance to the surgical margins between the two arms (1A and 1B).
* Study 2: to compare the anorectal functional outcome at 12 months after surgery or ileostomy closure between the two arms (2A and 2B). The anorectal function will be assessed by the scores of the validated Colorectal Functional Outcome Questionnaire (COREFO) and the validated scale LARS (Syndrome anterior resection of the rectum).

Secondary outcome measures:

* Study 1: to compare the duration of surgery, bleeding and need for surgical conversion between the two arms (1A and 1B). Another objectives are to compare the incidence of postoperative complications (measured by the Clavien-Dindo classification) and survival.
* Study 2: to compare the quality of life and anorectal functional outcomes at : 6, 12, 18 and 24 months after intervention (or ileostomy closure) between the two arms (2A and 2B). The anorectal function will be assessed by the validated COREFO questionnaire and the LARS scale. The quality of life will be assessed by the validated questionnaire of quality of life: SF-36. Another objective is to compare the incidence of postoperative complications assessed by the Clavien-Dindo classification and the incidence of anastomotic leakage.

Duration and follow up

Study 1: the expected study duration is 6'5 years.

Study 2: the expected duration of the study is 3'5 years.

The planned duration of follow up in the study 1 is 5 years, in the study 2 is 2 years.

Selection criteria

Inclusion Criteria:

Study 1:

* Patients with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer.
* Age ≥ 18 years
* Histology proven adenocarcinoma or adenoma with or without chemotherapy or neoadjuvant radiochemotherapy
* Any T, any N, M or any adenoma
* Attempt to R0 resection
* Signed informed consent by the patient and by the researcher
* Quality of Life Questionnaire completed

Study 2:

* Patients with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer with colorectal anastomosis.
* Age ≥ 18 years
* Histology proven adenocarcinoma or adenoma with or without chemotherapy or neoadjuvant radiochemotherapy
* Any T, any N, M or any adenoma
* Attempt to R0 resection
* Signed informed consent by the patient and by the researcher
* Quality of Life Questionnaire completed

Exclusion Criteria:

Study 1:

* Colorectal tumor with different histology to adenocarcinoma or adenoma
* History of colorectal cancer surgery different to the local excision
* Inflammatory bowel disease with pathologic confirmation
* Patients with psychiatric illness, addiction or disorder with inability to understand informed consent
* Inability to read or understand any of the languages of the informed consent and questionnaires (Catalan, spanish)
* Another synchronous malignancy
* Emergency Surgery
* Any patient that medical characteristics present an individual risk raised to be included and complete the study

Study 2:

* Patients who won't undergo colorectal anastomosis
* Colorectal tumor with different histology to adenocarcinoma or adenoma
* History of colorectal cancer surgery different to the local excision
* Inflammatory bowel disease with pathologic confirmation
* Patients with psychiatric illness, addiction or disorder with inability to understand informed consent
* Inability to read or understand any of the languages of the informed consent and questionnaires (Catalan, spanish)
* Another synchronous malignancy
* Emergency Surgery

ELIGIBILITY:
Inclusion Criteria:

Study 1:

* Patients with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer.
* Age ≥ 18 years
* Histology proven adenocarcinoma or adenoma with or without chemotherapy or neoadjuvant radiochemotherapy
* Any T, any N, M or any adenoma
* Attempt to R0 resection
* Signed informed consent by the patient and by the researcher
* Quality of Life Questionnaire completed

Study 2:

* Patients with colorectal cancer that will undergo laparoscopic left hemicolectomy or laparoscopic low anterior resection for rectal cancer with colorectal anastomosis.
* Age ≥ 18 years
* Histology proven adenocarcinoma or adenoma with or without chemotherapy or neoadjuvant radiochemotherapy
* Any T, any N, M or any adenoma
* Attempt to R0 resection
* Signed informed consent by the patient and by the researcher
* Quality of Life Questionnaire completed

Exclusion Criteria:

Study 1:

* Colorectal tumor with different histology to adenocarcinoma or adenoma
* History of colorectal cancer surgery different to the local excision
* Inflammatory bowel disease with pathologic confirmation
* Patients with psychiatric illness, addiction or disorder with inability to understand informed consent
* Inability to read or understand any of the languages of the informed consent and questionnaires (Catalan, spanish)
* Another synchronous malignancy
* Emergency Surgery
* Any patient that medical characteristics present an individual risk raised to be included and complete the study

Study 2:

* Patients who won't undergo colorectal anastomosis
* Colorectal tumor with different histology to adenocarcinoma or adenoma
* History of colorectal cancer surgery different to the local excision
* Inflammatory bowel disease with pathologic confirmation
* Patients with psychiatric illness, addiction or disorder with inability to understand informed consent
* Inability to read or understand any of the languages of the informed consent and questionnaires (Catalan, spanish)
* Another synchronous malignancy
* Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Total number of resected lymph nodes | 1 month
  Study 1:To compare the total number of resected lymph nodes between the two arms (1A and 1B).
Anorectal functional outcome at 12 months assessed by COREFO questionnaire | 12 months
  Study 2: to compare the anorectal functional outcome at 12 months after surgery or ileostomy closure between the two arms (2A and 2B). Assessed by the validated Colorectal Functional Outcome Questionnaire (COREFO)
Anorectal functional outcome at 12 months assessed by LARS scale | 12 months
  Study 2: to compare the anorectal functional outcome at 12 months after surgery or ileostomy closure between the two arms (2A and 2B). Assessed by the validated scale LARS (Syndrome anterior resection of the rectum).

SECONDARY OUTCOMES:
Intraoperative outcomes: duration of surgery | 1 day
  Study 1: to compare the duration of surgery measured in minutes between the two arms (1A and 1B).
Intraoperative outcomes: surgical bleeding | 1 day
  Study 1: to compare the surgical bleeding measured in ml between the two arms (1A and 1B).
Intraoperative outcomes: surgical conversion | 1 day
  Study 1: to compare the incidence of surgical conversion to laparotomy between the two arms (1A and 1B).
Postoperative complications | 90 days
  Study 1 and 2: Postoperative complications within 90 days after surgery (Clavien-Dindo classification).
Survival | 5 years
  Study 1: 5-year survival rate after surgery
Quality of life-SF questionnaire | 6, 12, 18 and 24 months after surgery
  Study 2: to compare the quality of life : 6, 12, 18 and 24 months after intervention (or ileostomy closure) between the two arms (2A and 2B). Assessed by the validated the validated questionnaire of quality of life: SF-36.
Anorectal functional outcome assessed by COREFO questionnaire | 6,18 and 24 months after surgery
  Study 2: to compare the anorectal functional outcomes at : 6, 18 and 24 months after intervention (or ileostomy closure) between the two arms (2A and 2B). Assessed by the validated Colorectal Functional Outcome Questionnaire (COREFO).
Postoperative complications and anastomotic leakage | 90 days after surgery
  Study 2: to compare the incidence of postoperative complications assessed by the Clavien-Dindo classification and the incidence of anastomotic leakage according to the classification of the International Group for Rectal Cancer Study.
Anorectal functional outcome assessed by LARS scale | 6,18 and 24 months after surgery
  to compare the anorectal functional outcomes at : 6, 18 and 24 months after intervention (or ileostomy closure) between the two arms (2A and 2B). Assessed by the validated scale LARS (Syndrome anterior resection of the rectum).
Distance to surgical margins | 1 month
  Study 1: To compare distance to surgical margins measured in mm between the group 1A and 1B

CONTACTS AND LOCATIONS:
Overall Officials: Pere Planellas Giné, MD-PhD, Principal Investigator — Colorectal Surgery Unit. Department of General and Digestive Surgery. University Hospital Dr. Josep Trueta of Girona
Locations (1):
- University Hospital Dr. Josep Trueta of Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Planellas P, Farres R, Cornejo L, Rodriguez-Hermosa JI, Pigem A, Timoteo A, Ortega N, Codina-Cazador A. Randomized clinical trial comparing side to end vs end to end techniques for colorectal anastomosis. Int J Surg. 2020 Nov;83:220-229. doi: 10.1016/j.ijsu.2020.09.039. Epub 2020 Oct 7. PMID 33038521